CLINICAL TRIAL: NCT01278732
Title: Central Blood Pressure Over 24 Hours (ABPM) and Left Ventricular Mas
Brief Title: Central Blood Pressure Over 24 Hours (ABPM) and Left Ventricular Mass
Status: Completed | Type: Observational
Sponsor: Klinikum Wels-Grieskirchen (Other)
Collaborators: Austrian Society of Hypertension (Unknown); European Regional Development Fund (Other); I.E.M. (Stolberg, Germany) (Unknown)
Responsible Party: Principal Investigator, Thomas Weber, PD Dr. Thomas Weber, Klinikum Wels-Grieskirchen
Other Study IDs: EK D-4-10
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Suspected Arterial Hypertension
Keywords: arterial hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- untreated persons with suspected hypertension
  Interventions: Other: no intervention performed

INTERVENTIONS:
Other: no intervention performed — no intervention is performed

SUMMARY:
The investigators aim to investigate whether central systolic blood pressure, as measured during regular 24 hour ambulatory blood pressure monitoring (ABPM), is a better predictor of left ventricular mass than peripheral systolic blood pressure during ABPM.

DETAILED DESCRIPTION:
It seems obvious that central blood pressures are pathophysiologically more relevant than peripheral blood pressures for the pathogenesis of cardiovascular disease: it is central systolic pressure (cSBP) against the heart ejects (afterload), and it is central pulse pressure (cPP) that distends the large elastic arteries. Indeed, cSBP and cPP have been associated more closely with left ventricular hypertrophy and carotid atherosclerosis as markers of hypertensive end-organ damage than brachial pressures in various populations. However, in these studies office blood pressure measurements have been used. As ABPM measurements per se show a closer association with hypertensive end-organ damage than office measurements, and as the investigators have recently developed and validated a novel algorithm (ARCSolver) to calculate central blood pressures from peripheral waveforms, the investigators speculate that cSBP measured during ABPM may be the best predictor of left ventricular mass.

ELIGIBILITY:
Inclusion Criteria:

> 18 years of age,

* no intake of antihypertensive medications
* should have an indication for ABPM (suspected arterial hypertension)

Exclusion Criteria:

* no written informed consent
* left ventricular hypertrophy due to other reasons than hypertension (hypertrophic cardiomyopathy, infiltrative cardiomyopathy, valvular heart disease, congenital heart disease)
* inability to provide adequate echocardiographic readings
* segmental contraction abnormalities of the left ventricle
* contraindications for ABPM (lymphedema both arms)
* other rhythm than stable sinus rhythm
* unstable clinical condition, including recent severe infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass (m-mode echocardiography) | measured within 4 weeks from ABPM

SECONDARY OUTCOMES:
urine albumine / creatinine ratio | measured within 2 weeks from ABPM but before antihypertensive treatment is started

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Weber, MD, associate professor, Principal Investigator — Cardiology Department, Klinikum Wels-Grieskirchen, Austria
Locations (10):
- Austria (2):
  - Cardiology Department, Klinikum Wels-Grieskirchen, Wels, Upper Austria
  - Cardiology Department, University of Graz, Graz
- Cardiology Department, University of Lübeck, Lübeck, Germany
- Sotiria Hospital 3rd Department of Internal Medicine, Athens, Greece
- Italy (3):
  - Department of Medical and Surgical Sciences, University of Brescia, Brescia
  - Clinica Medica, Hospitalo San Gerardo, Monza
  - Unit of Internal Medicine, Angiology and Arteriosclerosis, University of Perugia, Perugia
- Hospital de Sagunto, Port de Sagunt, Spain
- University of Basel, Basel, Switzerland
- Clinical pharmacology unit, University of Cambridge, Cambridge, United Kingdom

REFERENCES:
- [Derived] Weber T, Wassertheurer S, Schmidt-Trucksass A, Rodilla E, Ablasser C, Jankowski P, Lorenza Muiesan M, Giannattasio C, Mang C, Wilkinson I, Kellermair J, Hametner B, Pascual JM, Zweiker R, Czarnecka D, Paini A, Salvetti M, Maloberti A, McEniery C. Relationship Between 24-Hour Ambulatory Central Systolic Blood Pressure and Left Ventricular Mass: A Prospective Multicenter Study. Hypertension. 2017 Dec;70(6):1157-1164. doi: 10.1161/HYPERTENSIONAHA.117.09917. Epub 2017 Oct 23. PMID 29061725